CLINICAL TRIAL: NCT02922036
Title: Stimulation Of the Left Ventricular Endocardium for Cardiac Resynchronization Therapy in Non-Responders, Previously Untreatable and High Risk Upgrade Patients (SOLVE CRT)
Brief Title: Cardiac Resynchronization Therapy in Previously Untreatable and High Risk Upgrade Patients
Acronym: SOLVE-CRT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EBR Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CSP-03035
Record Dates: First submitted 2016-09-27; First posted 2016-10-03 (Estimated); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Masking Description: One part of the study was randomized. The final part of the study was single-arm, open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): WiSE System therapy ON with Guideline Directed Medical Therapy
  Interventions: Device: WiSE System

INTERVENTIONS:
Device: WiSE System — The WiSE System is an implantable cardiac system to provide LV pacing stimulation in conjunction with a co-implanted system that provides right ventricular stimulation.

SUMMARY:
This study is a prospective, multi-center, pivotal trial to study the safety and efficacy of the WiSE-CRT System for Cardiac Re-synchronization Therapy.

DETAILED DESCRIPTION:
The WiSE-CRT System is an implantable cardiac pacing system capable of delivering pacing energy to the left ventricle of the heart without using a pacing lead.

ELIGIBILITY:
Inclusion/Exclusion:

Inclusion Criteria

1. Patient with a class I or IIa (1) or (2) indication for implantation of a CRT-D device according to current available guidelines (with additional QRS criteria on Class IIa (1)):

   1. Class I: NYHA II, III, IV, EF ≤ 35%, LBBB, QRS ≥ 150ms
   2. Class IIa (1): NYHA II, III, IV, EF≤ 35%, LBBB, QRS ≥ 130 to < 150ms
   3. Class IIa (2): NYHA II, III, IV, EF≤ 35%, non-LBBB, QRS ≥ 150ms
2. Patient is a:

   1. 'Non-responder' [Not Enrolling]: Patients who have a CRT system that is functional and despite an adequate trial of Guideline Directed Medical Therapy (GDMT) and attempts at optimal device programming the patient has not responded to therapy for a minimum of 6 months. Non-response is defined as:

      * EF has remained unchanged or worsened (defined as < 5% increase since implant), and
      * The patient's clinical status based in the totality of available clinical evidence (such as NYHA Class, exercise tolerance, QOL, or global assessment) has remained unchanged or worsened, as determined by the local Site Enrollment Committee

      OR
   2. 'Previously Untreatable': Patients who have a full or partial CRT system, who meet general inclusion criteria and are deemed as 'previously untreatable' for one of the following reasons:

   i. Patients in whom CS lead implantation for CRT has failed
   * CS lead implant was attempted but abandoned due any of the following: difficult CS access or anatomy, inadequate lead location, inadequate pacing thresholds, persistent phrenic nerve pacing, or other procedural challenges

   ii. CS lead implanted but has been programmed OFF
   * LV lead that was implanted but not operational includes patients in whom the LV lead is inoperative or programmed off due to improper function such as high threshold, non-capture, phrenic nerve pacing, lead failure, lead dislodgement, or sub-optimal LV lead location

   OR

   c. 'High Risk Upgrade:

   Patients who have a relative contraindication to CS lead implant, due to:
   * venous occlusion or lesion precluding implant
   * pocket infection risk (at co-implanted device site)
   * considered high risk for CS implant due to co-morbidities
3. Patients on a stable Guideline Directed Medical Therapy (GDMT)
4. Patient must be 18 years old or over
5. Patient has signed and dated informed consent
6. Patient has suitable anatomy for implant of the WiSE CRT System (e.g. adequate acoustic window, LV wall thickness in target implant area ≥ 5 mm, absence of LV wall structural abnormalities which may preclude implant)

Exclusion Criteria

Patients who meet any one of these criteria will be excluded from the investigation:

1. Pure RBBB
2. LVEDD ≥ 8cm
3. Non-ambulatory or unstable NYHA class IV
4. Contraindication to heparin, chronic anticoagulants or antiplatelet agents
5. Triple anticoagulant patients who cannot tolerate peri-procedural stopping of anticoagulation therapy
6. Attempted device implant (pacemaker, ICD, CRT, LV lead) or successful co-implant within prior 30 days.
7. Patients with planned or expected lithotripsy treatment post implant
8. Life expectancy of < 12 months
9. Chronic hemodialysis
10. Stage 4 or 5 renal dysfunction defined as eGFR < 30
11. Grade 4 mitral valve regurgitation
12. Noncardiac implanted electrical stimulation therapy devices
13. Patients with a prosthetic aortic valve in which the electrode cannot be implanted via a transseptal approach
14. Patients with a prosthetic mitral valve in which the electrode cannot be implanted via a retrograde aortic approach
15. Unstable angina, acute MI, CABG, or PTCA within the past 1 month
16. Correctable valvular disease that is the primary cause of heart failure
17. Recent CVA or TIA (within the previous 3 months)
18. Patients with a history of paroxysmal or persistent atrial fibrillation/flutter are excluded if they have had a documented AF episode > 30 min or a cardioversion in the past 1 month.
19. Patients with permanent AF are excluded if they have intact AV node conduction (RV pacing <95%)
20. Already included in another clinical study that could confound the results of this study
21. Pregnancy
22. Known drug or alcohol addiction or abuse
23. Moderate or severe aortic stenosis
24. Subject unable to attend follow-up at the investigative center or unable, for physical or mental reasons, or to comply with the trial's procedures
25. For Part II Randomized patients only, those who will not tolerate being randomized to the Control Group for 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary Safety | 6 Months
  Freedom from Procedure and Device System related Type 1 Complications
Primary Efficacy 1 | 6 Months
  Mean relative % change in Left Ventricular End Systolic Volume (LVESV) baseline to 6 Months.

SECONDARY OUTCOMES:
Secondary Efficacy 1 | 6 Months
  Electrode Acoustic Pacing Capture Threshold (APCT) measured at the 6-month follow-up post-implant visit
Secondary Efficacy 2 | 6 Months
  Electrode Acoustic Pacing Capture Threshold Stability (APCT Stability) measured from pre-discharge through the 6-month follow-up post-implant visit
Secondary Efficacy 3 | 6 months
  % Bi-ventricular pacing at 6 months
Secondary Efficacy 4 | 6 months
  EF responder analysis for ≥ 5% absolute increase from baseline to 6 months.
Secondary Efficacy 5 | 6 months
  KCCQ responder analysis for ≥ 5 points absolute increase from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jagmeet Singh, MD, PhD, Principal Investigator — Massachusetts General Hospital; Mary N Walsh, MD, MACC, Principal Investigator — St. Vincent Heart Center
Locations (68):
- United States (43):
  - Heart Center Research, Huntsville, Alabama
  - University of California, San Diego, La Jolla, California
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - St. Vincent's Healthcare, Jacksonville, Florida
  - Watson Clinic, Lakeland, Florida
  - Naples Community Hospital, Naples, Florida
  - Northside Hospital and Heart Institute, St. Petersburg, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory Healthcare, Atlanta, Georgia
  - Prairie Heart, Springfield, Illinois
  - St. Vincent's Hospital and Healthcare Center, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Saint Luke's Health System Kansas City, Kansas City, Kansas
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Ochsner Medical Center - Baton Rouge, Baton Rouge, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Michigan Heart, Canton, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Hazel Park, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Methodist Physicians Clinic Heart Consultants, Omaha, Nebraska
  - Rutgers University, New Brunswick, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Weill Cornell Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - PeaceHealth, Springfield, Oregon
  - Penn State Health, Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Heart and Vascular Institute, Pittsburgh, Pennsylvania
  - MUSC Gazes Research Institute, Charleston, South Carolina
  - Stern Cardiovascular Center, Germantown, Tennessee
  - Texas Heart Institute, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Houston Methodist, Sugar Land, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Healthcare, Norfolk, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (10):
  - Canberra Hospital, Garran, Australian Capital Territory
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Heart, Clayton, Victoria
  - Royal Melbourne Hospital / Royal Hobart Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Perth, Western Australia
  - Royal Prince Alfred Hospital, Camperdown
- France (3):
  - CHU Grenoble - Hopital Michallon Service de Cardiologie, Grenoble
  - Centre Cardiologique du Nord, Paris
  - CHU-Hopital Pontchaillou, Rennes
- Germany (3):
  - Immanuel Klinikum Bernau - Herzzentrum Brandenburg, Bernau
  - Universitätsklinikum Erlangen, Erlangen
  - Universitäres Herzzentrum Hamburg (UKE Hamburg) GmbH (UHZ), Hamburg
- Italy (2):
  - Policlinico S. Orsola, Bologna
  - Ospedale San Gerardo, Monza
- Isala Hartcentrum, Zwolle, Netherlands
- United Kingdom (6):
  - Liverpool Heart and Chest Hospital, Liverpool
  - Barts Heart Centre, London
  - St. Thomas Hospital, London
  - Manchester Heart Centre, Manchester
  - James Cook University Hospital, Middlesbrough
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh JP, Abraham WT, Auricchio A, Delnoy PP, Gold M, Reddy VY, Sanders P, Lindenfeld J, Rinaldi CA. Design and rationale for the Stimulation Of the Left Ventricular Endocardium for Cardiac Resynchronization Therapy in non-responders and previously untreatable patients (SOLVE-CRT) trial. Am Heart J. 2019 Nov;217:13-22. doi: 10.1016/j.ahj.2019.04.002. Epub 2019 Apr 9. PMID 31472360
- See also: Leadless Ultrasound-Based Cardiac Resynchronization System in Heart Failure — https://pmc.ncbi.nlm.nih.gov/articles/pmid/39083254/